CLINICAL TRIAL: NCT05563090
Title: Investigating the Syndrome Differentiation of Diabetic and Pre-diabetic Patients in Singapore Using Digitalized TCM Diagnostic Tools: an Observational Study
Brief Title: Investigating the Syndrome Differentiation of Diabetic and Pre-diabetic Using Digitalized TCM Diagnostic Tools
Status: Completed | Type: Observational
Sponsor: Singapore Chung Hwa Medical Institution (Other)
Collaborators: Ministry of Health, Singapore (Other Government)
Responsible Party: Sponsor
Other Study IDs: SCHMI-2022-001
Record Dates: First submitted 2022-09-25; First posted 2022-10-03 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2023-12

CONDITIONS: Diabete Mellitus; Pre-diabetes; Healthy; Hypertension; Dyslipidemia Associated With Type II Diabetes Mellitus
Keywords: Diabetes Mellitus; Type II diabetes; Pre-diabetes; Healthy subjects; hypertension; dyslipidemia; TCM; TCM diagnosis; Pulse diagnosis; Tongue diagnosis
MeSH Terms: conditions — Diabetes Mellitus; Glucose Intolerance; Hypertension; Diabetes Mellitus, Type 2; Dyslipidemias

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (5):
- 0HEA: Healthy or sub-healthy subject without clinically diagnosed chronic conditions such as diabetes, hypertension or dyslipidemia
  Interventions: Other: Questionnaires+Tongue diagnosis+Pulse diagnosis
- 1PRE: Prediabetes with IFG of FPG 6.1-6.9 mmol/L, and/or IGT with 2hPG of 7.8-11.0 mmol/L
  Interventions: Other: Questionnaires+Tongue diagnosis+Pulse diagnosis
- 2DIA: Diabetes with FPG of ≥ 7.0 mmol/L, 2hPG of ≥ 11.1mmol, or HbA1c of > 6.5%
  Interventions: Other: Questionnaires+Tongue diagnosis+Pulse diagnosis
- 3PREHD: Prediabetes with hypertension and dyslipidemia
  Interventions: Other: Questionnaires+Tongue diagnosis+Pulse diagnosis
- 4DIAHD: Diabetes with hypertension and dyslipidemia
  Interventions: Other: Questionnaires+Tongue diagnosis+Pulse diagnosis

INTERVENTIONS:
Other: Questionnaires+Tongue diagnosis+Pulse diagnosis — Each subject will undergo questionnaires, tongue and pulse diagnosis using modern diagnostic tools

SUMMARY:
The investigators aim to objectively identify the Traditional Chinese Medicine (TCM) syndrome differentiation of type II diabetic and prediabetic patients in Singapore through modern technologies thereby potentially increasing the accuracy of identification, diagnosis, and prevention of diabetes and prediabetes through a system of targeted treatment. This observational study integrates the concept of TCM diagnostic methods with modern tools aim to provide an objective view on the syndrome differentiation of diabetic and prediabetic patients in Singapore and hence provide a guideline in the treatment options targeted specifically at Singaporeans demographic.

A total of 250 subjects with 50 allocated in each group will be recruited to ensure a sufficient sample size for statistical analysis of the diabetic and prediabetic syndrome differentiation. Subjects aged 21-65 years old, of either gender, with no limitations on race, and is diagnosed with either diabetes (FPG ≥ 7.0 mmol/L, or 2hPG ≥ 11.1mmol) or prediabetes (IFG of FPG 6.1-6.9 mmol/L, and/or IGT with 2hPG of 7.8-11.0 mmol/L) will be included.

Subjective and objective assessments through health evaluation, Physical Activity Questionnaire and Sugar Intake, Constitution in Chinese Medicine Questionnaire, radial pulse diagnosis and tongue diagnosis will be performed for each subject in a single visit. Statistical analysis of assessments will be conducted using unpaired t-test with significance level of p<0.05. Statistical software SPSS 15.0 (SPSS Inc.) will be used for the analysis.

DETAILED DESCRIPTION:
Singapore's age-adjusted comparative prevalence of diabetes is at 5.5% in 2019 down from 10.2% in 2010, whereas the global average is at 8.3%. However, approximately 640,000 Singapore citizens 18 years and above are diagnosed with diabetes, and around 650,000 citizens are prediabetic.

The investigators aim to objectively identify the Traditional Chinese Medicine (TCM) syndrome differentiation of type II diabetic and prediabetic patients in Singapore through modern technologies thereby potentially increasing the accuracy of identification, diagnosis, and prevention of diabetes and prediabetes through a system of targeted treatment.

The investigators hypothesize that the TCM syndrome differentiation of 'xiao-ke' in Singapore is different from that of the ones defined in TCM Internal Medicine, which is based on China demographics.

This observational study integrates the concept of TCM diagnostic methods with modern tools aim to provide an objective view on the syndrome differentiation of diabetic and prediabetic patients in Singapore and hence provide a guideline in the treatment options targeted specifically at Singaporeans demographic.

The investigators will attempt to recruit a total of 250 subjects with 50 allocated in each group to ensure a sufficient sample size for statistical analysis of the diabetic and prediabetic syndrome differentiation. Subjects aged 21-75 years old, of either gender, with no limitations on race, and is diagnosed with either diabetes (FPG ≥ 7.0 mmol/L, or 2hPG ≥ 11.1mmol) or prediabetes (IFG of FPG 6.1-6.9 mmol/L, and/or IGT with 2hPG of 7.8-11.0 mmol/L) will be included.

Subjective and objective assessments through health evaluation, Physical Activity Questionnaire and Sugar Intake, Constitution in Chinese Medicine Questionnaire, radial pulse diagnosis and tongue diagnosis will be performed for each subject in a single visit. Statistical analysis of assessments will be conducted using unpaired t-test with significance level of p<0.05. Statistical software SPSS 15.0 (SPSS Inc.) will be used for the analysis.

ELIGIBILITY:
Inclusion Criteria:

* Aged 21-75 years old, inclusive;
* Clinically diagnosed with one of the following:

  1. Type II Diabetes Mellitus with or without hypertension and dyslipidemia
  2. Prediabetes with or without hypertension and dyslipidemia
  3. Healthy or sub-healthy subject without clinically diagnosed chronic conditions such as diabetes, hypertension or dyslipidemia

Exclusion Criteria:

* Subjects diagnosed with Gestational Diabetes
* Subjects who are pregnant or lactating
* Subjects with chronic heart failure, history of carcinomas with treatment of chemotherapy/radiotherapy, psychological, or psychiatric disorders
* Subjects with heart diseases and transplanted devices such as pacemakers;
* Subjects with acute infections such as upper respiratory infections, acute gastroenteritis, or urinary tract infections;
* Subjects unable to undergo evaluation with the pulse sphygmograph, tongue detection or complete the questionnaire;
* Subjects with communication disorders
* Subjects with gastroenterology diseases or are diagnosed with 'spleen and stomach deficiency' (脾胃虚弱)
* Subjects undergoing TCM treatment for diabetes or pre-diabetes within 1 week

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The subjects need to be at 21-75 years old, of either gender, with no limitations on race, and is clinically diagnosed by Western medical doctors with either diabetes (FPG of ≥ 7.0 mmol/L, 2hPG of ≥ 11.1mmol, or HbA1c of > 6.5%) or prediabetes (IFG of FPG 6.1-6.9 mmol/L, and/or IGT with 2hPG of 7.8-11.0 mmol/L). Healthy or sub-healthy subjects without any significant health related issues, eg. clinically diagnosed chronic conditions such as diabetes, hypertension or dyslipidemia, will be recruited as the control group. The health evaluation form (Annex 1) will be used to verify that these healthy subjects (1) do not have any family history of diabetes, and (2) do not have unusual high fasting blood glucose detected within one year.
Sampling Method: Non-Probability Sample
Enrollment: 171 (Actual)
Dates: Start 2022-09-17 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2025-04-01 (Actual)

PRIMARY OUTCOMES:
The Constitution in Chinese Medicine Questionnaire (CCMQ) | One-time assessment within 30mins before undergoing the tongue and pulse diagnosis.
  The CCMQ, published by the China Association of Chinese Medicine in 2009, will be adopted to assess the body constitution of each subjects based on TCM principles [26]. Refer to Annex 3.
  There are nine different types of body constitution, including (a) Normality; (b) Qi deficiency; (c) Yin deficiency; (d) Yang deficiency; (e) Phlegm-dampness; (f) Damp-heat; (g) Blood stasis; (h) Qi depressed; (i) Inherited special constitution.
  Each subject will answer seven to eight questions in each category. The scoring algorithm indicates the likelihood of a specific type of body constitution with a higher score.
Physical Activity Questionnaire and sugar intake | One-time assessment within 30mins before undergoing the tongue and pulse diagnosis.
  Level of physical activity related to the last three months will be recorded through the Physical Activity Questionnaire. Sugar intake includes sweet or carbonated drinks, desserts like chocolates and cakes, 0 - 2, 3 - 6, or more than 7 times a week will also be recorded. Refer to Annex 2.
  This will help to identify the risk factors involved and identify the correlation between the body constitutions and various types of 'xiao-ke' based on TCM syndrome differentiation.
Pulse sphygmograph | One-time assessment within 30mins after undergoing the questionnaires
  The Asia Plus Pen Pulse Analysis System Model PPAS-93 (Asia Plus Bio Tech Co., Ltd, Taiwan) would be used in the identification of RPPW of the subjects in this study.
  The Asia Plus Pen Pulse Analysis System Model PPAS-93 (Figure 11) is a noninvasive device that consist of a high precision pressure sensor pen and a pulse analyzer. The 3D pulse detector is a handheld pen that digitalizes the biological signal of RPPW and provides a graphical analysis. The electronic device contains a high precision pressure sensor, a filter, an amplifier, and a signal recording card connected to signal analysis software. The frequency response is 0.1-50 Hz, and the sampling rate is 3000 Hz.
Tongue imaging device | One-time assessment within 30mins after undergoing the questionnaires
  China Artificial Intelligence Health Status Identification System Model Number YZKJ-SMZY-1AI (Figure 12) will be used in the imaging and analysis of the subject's tongue.
  The noninvasive device captures the image of the tongue through an inbuilt camera supported by LED lights within the device. A monitor that is connected to the imaging device would provide a live video feedback on the positioning of the tongue. The images of the subjects' face, tongue, and sublingual collaterals will then be compared and analyzed for the similarities against standard images of tongue analysis using an artificial intelligence system.

SECONDARY OUTCOMES:
Health Evaluation - Age | One-time assessment within 30mins before undergoing the tongue and pulse diagnosis.
  Demographic information eg age in years will be collected.
Health Evaluation - Gender | One-time assessment within 30mins before undergoing the tongue and pulse diagnosis.
  Demographic information eg gender will be collected.
Health Evaluation - Weight | One-time assessment within 30mins before undergoing the tongue and pulse diagnosis.
  Weight in kilogram will be recorded
Health Evaluation - Height | One-time assessment within 30mins before undergoing the tongue and pulse diagnosis.
  Height in meters will be recorded
Health Evaluation - BMI | One-time assessment within 30mins before undergoing the tongue and pulse diagnosis.
  Weight in kilogram and height in meters will be aggregated to derive the BMI in kg/m^2.
Health Evaluation - blood sugar level | One-time assessment within 30mins before undergoing the tongue and pulse diagnosis.
  Blood glucose in fasting, 2hPG or HbA1c (in mmol/L) results if available in patient's regular blood test report
Health Evaluation - Vital signs | One-time assessment within 30mins before undergoing the tongue and pulse diagnosis.
  Vital signs including systolic blood pressure, diastolic blood pressure in mmHg
Health Evaluation - Radial pulse rate | One-time assessment within 30mins before undergoing the tongue and pulse diagnosis.
  Vital signs including radial pulse rate (bpm)
Health Evaluation - Medications | One-time assessment within 30mins before undergoing the tongue and pulse diagnosis.
  Western and Chinese medications and nutritional supplements consumed by the subjects will be recorded to identify possible intervention and correlation towards TCM syndrome differentiation.
Health Evaluation - Existing symptoms | One-time assessment within 30mins before undergoing the tongue and pulse diagnosis.
  The existing symptoms of subjects will be recorded to identify the possible correlation towards TCM syndrome differentiation.

CONTACTS AND LOCATIONS:
Locations (1):
- Singapore Chung Hwa Medical Institution, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ng HP, Chong SY, Li YH, Goh TH, Pang KY, Pereira MJ, Huang CM. Objective Analysis of Traditional Chinese Medicine Syndrome Differentiation of Patients With Diabetes and Prediabetes: Protocol for a Nonrandomized, Exploratory, Observational Case-Control Study Using Digitalized Traditional Chinese Medicine Diagnostic Tools. JMIR Res Protoc. 2024 Sep 12;13:e56024. doi: 10.2196/56024. PMID 39265161